CLINICAL TRIAL: NCT07162935
Title: Addiction Potential, Flavoring Content, and Substitutability of Concept Flavored Cigarillos
Brief Title: Cigar Legislation and Regulation in Tobacco for the Young (Project CLARITY)
Acronym: Clarity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Clarity; R01DA062632-01 (NIH)
Record Dates: First submitted 2025-09-02; First posted 2025-09-09 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Cigar Smoking; Tobacco Use
MeSH Terms: conditions — Cigar Smoking; Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Concept flavor (Experimental): Participants will be randomized to smoke one of the three assigned concept flavored cigarillos
  Interventions: Other: Cigarillo brand 1; Other: Cigarillo brand 2; Other: Cigarillo brand 3
- Characterizing flavor (Experimental): Participants will be randomized to smoke one of the three assigned characterizing flavored cigarillos
  Interventions: Other: Cigarillo brand 1; Other: Cigarillo brand 2; Other: Cigarillo brand 3
- Tobacco flavor (Experimental): Participants will be randomized to smoke a tobacco flavored cigarillo
  Interventions: Other: Cigarillo brand 1; Other: Cigarillo brand 2; Other: Cigarillo brand 3

INTERVENTIONS:
Other: Cigarillo brand 1 — Participants will be assessed on puffing behavior, subjective effects, and exhaled carbon monoxide when assigned to using one of three cigarillo brands. Additives and ingredients of the cigarillo used will also be assessed
Other: Cigarillo brand 2 — Participants will be assessed on puffing behavior, subjective effects, and exhaled carbon monoxide when assigned to using one of three cigarillo brands. Additives and ingredients of the cigarillo used will also be assessed
Other: Cigarillo brand 3 — Participants will be assessed on puffing behavior, subjective effects, and exhaled carbon monoxide when assigned to using one of three cigarillo brands. Additives and ingredients of the cigarillo used will also be assessed

SUMMARY:
This clinical trial will recruit young adults who currently use cigarillos and examine the smoking behavior and perceptions of different flavored cigarillos, product ingredients/additives impacting these perceptions, and simulated tobacco use outcomes (quitting, switching) in various policy scenarios where different types of flavors are available on the market.

DETAILED DESCRIPTION:
This clinical trial will isolate the unique effects of concept descriptors on increased cigarillo use and appeal among experienced young adult cigarillo users. The study will seek to determine the addiction potential of concept flavored cigarillos by examining associations of cigarillo flavor type (concept, characterizing, tobacco) and cigarillo flavoring additives/ingredients to complementary measures of product appeal: subjective effects (e.g., satisfaction, reward, taste), actual smoking behavior (e.g., number of puffs), and simulated cigarillo purchasing, other tobacco product substitution, or quitting under different flavor ban scenarios via an Experimental Tobacco Marketplace (ETM).

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 to 24
2. Report past 30-day use of a cigarillo
3. Ability to read English at least an 8th grade level
4. No immediate plans to quit using tobacco
5. At least 1 prior experience with a flavored tobacco product
6. U.S. Citizen or permanent resident of the United States.

Exclusion Criteria:

1. Current use of smoking cessation pharmacotherapy or nicotine replacement therapy;
2. Pregnant, planning to become pregnant, or currently breastfeeding;
3. Past or current clinically significant heart disease or hypertension, or other smoking-related disease that could preclude successful study completion;
4. Inability to abstain from nicotine/tobacco products for at least 12 hours
5. Unwillingness to use the research cigarillos in the lab

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2030-03-02 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Puff number | From enrollment to the end of the final smoking visit, approximately 2 weeks
  Number of cigarillo puffs
Subjective reward from smoking | From enrollment to the end of the final smoking visit, approximately 2 weeks
  Self-reported reward from cigarillo smoking from a questionnaire. This scale has 5 questions with response options ranging from 1 - not at all to 7 - extremely. The score is averaged across the number of items. Higher ratings indicate greater psychological reward

CONTACTS AND LOCATIONS:
Overall Officials: Amy Cohn, OhD, Principal Investigator — University of Oklahoma Health Sciences
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Data that are determined to be private (name, address, email address) will be provided under a restricted data use contract to those who demonstrate a valid need and meet the conditions of use
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The investigative team will meet the data submission and release timeframes specified by the funding agency and policies, as described on NIH's data sharing webpage.